CLINICAL TRIAL: NCT03058900
Title: Efficacy and Safety of Fecal Microbiota Transplantation (FMT) in Patients With Peripheral Psoriatic Arthritis: a 6-month, Double-Blind, Randomized, Placebo-Controlled Trial
Brief Title: Efficacy and Safety of Fecal Microbiota Transplantation in Peripheral Psoriatic Arthritis
Acronym: FLORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other); The Danish Rheumatism Association (Other); Odense Patient Data Explorative Network (Other); The Psoriasis Association, Denmark (Unknown); Manufacturer Vilhelm Pedersen Foundation (Other); The Danish Regions (Medicinpuljen) (Unknown)
Responsible Party: Principal Investigator, Torkell Ellingsen, Clinical professor/Head of research and chief consultant MD PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OUH-DC-FLORA-01
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Psoriatic Arthritis
Keywords: Fecal Microbiota Transplantation; FMT; Randomized Controlled Trial; Intestinal microbiome; RCT; Faecal microbiota transplantation
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Fecal Microbiota Transplantation; Sodium Chloride; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation (FMT) (Experimental)
  Interventions: Drug: Fecal microbiota transplantation (FMT); Drug: Methotrexate (MTX)
- Placebo (saline) (Sham Comparator)
  Interventions: Other: Drug: Placebo (saline); Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Fecal microbiota transplantation (FMT) — One fecal microbiota transplantation is performed at baseline using gastroscopic guidance. The transplant consists of 50 g feces obtained from a healthy non-related donor. The donor feces is suspended into NaCl (0.9%) and glycerol (10%), and will be stored at minus 80 degrees celsius until use. The total volume of the suspension is 250 mL and its temperature will be 37 degrees celsius when infused into the small intestine of the recipient.
  Arms: Fecal microbiota transplantation (FMT)
Other: Drug: Placebo (saline) — One identical appearing sham procedure is performed at baseline using gastroscopic guidance. 250 mL saline (NaCl 0.9%) is infused into the small intestine of the recipient.
  Arms: Placebo (saline)
Drug: Methotrexate (MTX) — Weekly methotrexate in maximum tolerable dosis

SUMMARY:
An abnormal intestinal microbiota may be the mediator of the common inflammatory pathways seen in psoriatic arthritis. This study will explore clinical aspects associated with modifying the intestinal microbiota by infusing fecal donor microbiota into the small intestine of psoriatic arthritis patients with a minimum of three swollen joints despite at least three months of methotrexate treatment.

DETAILED DESCRIPTION:
Recent years have seen growing recognition of the complexity of the role of the microbiota in shaping the immune system and its potential effects for health and disease. In particular, the gut bacteria composition has been associated with the pathogenesis of autoimmune and inflammatory diseases. Intriguingly, presence of intestinal inflammation in psoriatic arthritis (PsA) patients has been documented in several studies. Also, in genetically predisposed patients reactive arthritis, which share some of the clinical manifestations of PsA, can be triggered by certain types of bacterial gut infections. Furthermore, a recent study has reported that several intestinal bacteria including Akkermansia and Ruminoccocus, which are known to play an important role in maintaining gut homeostasis, were practically absent in PsA patients. Mechanisms through which the microbiota may be involved in the pathogenesis of PsA include an abnormal activation of the gut-associated lymphoid tissue (GALT) and/or an altered mucosal permeability thus compromising the capacity of the intestine to provide adequate containment of luminal microorganisms and molecules.

By conducting a double-blinded, randomized, placebo-controlled trial of a non-related donor fecal microbiota transplantation (FMT) infused into the small intestine, this study will reveal whether FMT is more effective than an identically appearing placebo (saline) in reducing disease activity in psoriatic arthritis patients presenting with a minimum of three swollen joints despite at least three months of methotrexate treatment (maximal tolerable dosis ≥ 15 mg/week). All patients will throughout the study continue their individual treatment with weekly methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psoriatic arthritis according to the Classification Criteria for Psoriatic Arthritis (CASPAR criteria).
* Presence of active peripheral psoriatic arthritis defined as ≥ 3 swollen joints.
* Methotrexate (≥ 15mg/week (maximal tolerable dosage)) for a minimum of 3 months prior to study inclusion.

Exclusion Criteria:

* Other inflammatory rheumatic diseases than PsA.
* Current axial disease activity or severe peripheral joint activity demanding immediate change of treatment or contraindicating placebo treatment for 6 months.
* History of severe MTX toxicity or allergic reactions.
* Current biological treatment and biological treatment within the last 6 months.
* Inflammatory bowel disease, celiac disease, food allergy, or other intestinal diseases.
* Current cancer or severe chronic infections.
* Pregnant or breastfeeding women.
* Systemic and/or local intra-articular or peritendinous steroid injections within 3 months of inclusion.
* Non-MTX DMARD treatment within three months of inclusion.
* Antibiotics within 3 months of inclusion.
* Not wishing to participate or unsuited for project evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 6 months (+/- 14 days)
  Proportion of patients in each group who experience treatment failure according to shared decision making between patient and rheumatologist defined as at least one of the following:
  * Need for more than 1 intra-articular glucocorticoid injection due to disease activity.
  * Need for change to other conventional DMARDs (at the moment oral leflunomide, sulfasalazin or ciclosporin) according to the updated Danish guideline treatment due to disease activity.
  * Need for biologic treatment according to the updated Danish guideline treatment due to severe disease activity.

SECONDARY OUTCOMES:
The Short Health Assessment Questionnaire (2-page HAQ) | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Change from baseline in the Short Health Assessment Questionnaire (2-page HAQ).
The Dermatology Life Quality Index (DLQI) Questionnaire | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Change from baseline in the Dermatology Life Quality Index (DLQI).
Patient Reported Gastrointestinal Side Effects | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Change from baseline in gastrointestinal symptoms.
Patient Reported Other Side Effects | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Change from baseline in other (non-gastrointestinal) symptoms.
The American College of Rheumatology (ACR) Response Criteria | Baseline, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Proportion of patients in each group achieving
  * ACR20 response criteria
  * ACR50 response criteria
  * ACR70 response criteria
  A patient will be considered as improved according to the ACR20/50/70 response criteria if she/he has at least 20/50/70% improvement in the two following measures: Tender joint count (68) and swollen joint count (66), and at least 3 of the following 5 measures: Patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ) score, acute phase reactant (CRP).
The Psoriatic Arthritis Response Criteria (PsARC) | Baseline, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Proportion of patients in each group achieving PsARC response criteria. A patient will be considered as improved according to the PsARC response criteria if she/he has an improvement in either joint swelling or tenderness, and in any of 4 other measures: Patient global assessment of articular disease; physician global assessment of articular disease; joint pain or tenderness; joint swelling.
The Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index | Baseline, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Change from baseline in SPARCC Enthesitis Index in the subset of patients who have enthesitis at baseline.
The Psoriasis Area Severity Index (PASI) | Baseline, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Change from baseline in the Psoriasis Area Severity Index (PASI) in the subset of patients who have psoriasis at baseline.
Dactylitis | Baseline, 3 months (+/- 7 days), 6 months (+/- 14 days)
  Change from baseline in the number of digits affected with dactylitis in the subset of patients who have dactylitis at baseline.
Number of Adverse Events | 6 months (+/- 14 days)
  Number of adverse events in each group.
Number of Patients with Adverse Events | 6 months (+/- 14 days)
  Number of patients with at least one adverse event in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Torkell J. Ellingsen, Prof PhD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Dept. of Rheumatology at Odense University Hospital, Odense
  - Diagnostic Centre at Silkeborg Regional Hospital, Silkeborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coates LC, Conaghan PG, Emery P, Green MJ, Ibrahim G, MacIver H, Helliwell PS. Sensitivity and specificity of the classification of psoriatic arthritis criteria in early psoriatic arthritis. Arthritis Rheum. 2012 Oct;64(10):3150-5. doi: 10.1002/art.34536. PMID 22576997
- [Background] Taylor W, Gladman D, Helliwell P, Marchesoni A, Mease P, Mielants H; CASPAR Study Group. Classification criteria for psoriatic arthritis: development of new criteria from a large international study. Arthritis Rheum. 2006 Aug;54(8):2665-73. doi: 10.1002/art.21972. PMID 16871531
- [Background] Kingsley GH, Kowalczyk A, Taylor H, Ibrahim F, Packham JC, McHugh NJ, Mulherin DM, Kitas GD, Chakravarty K, Tom BD, O'Keeffe AG, Maddison PJ, Scott DL. A randomized placebo-controlled trial of methotrexate in psoriatic arthritis. Rheumatology (Oxford). 2012 Aug;51(8):1368-77. doi: 10.1093/rheumatology/kes001. Epub 2012 Feb 17. PMID 22344575
- [Background] Statnikov A, Alekseyenko AV, Li Z, Henaff M, Perez-Perez GI, Blaser MJ, Aliferis CF. Microbiomic signatures of psoriasis: feasibility and methodology comparison. Sci Rep. 2013;3:2620. doi: 10.1038/srep02620. PMID 24018484
- [Background] Eppinga H, Konstantinov SR, Peppelenbosch MP, Thio HB. The microbiome and psoriatic arthritis. Curr Rheumatol Rep. 2014 Mar;16(3):407. doi: 10.1007/s11926-013-0407-2. PMID 24474190
- [Background] Jacques P, Elewaut D. Joint expedition: linking gut inflammation to arthritis. Mucosal Immunol. 2008 Sep;1(5):364-71. doi: 10.1038/mi.2008.24. Epub 2008 Jul 9. PMID 19079200
- [Background] Scher JU, Sczesnak A, Longman RS, Segata N, Ubeda C, Bielski C, Rostron T, Cerundolo V, Pamer EG, Abramson SB, Huttenhower C, Littman DR. Expansion of intestinal Prevotella copri correlates with enhanced susceptibility to arthritis. Elife. 2013 Nov 5;2:e01202. doi: 10.7554/eLife.01202. PMID 24192039
- [Background] Brusca SB, Abramson SB, Scher JU. Microbiome and mucosal inflammation as extra-articular triggers for rheumatoid arthritis and autoimmunity. Curr Opin Rheumatol. 2014 Jan;26(1):101-7. doi: 10.1097/BOR.0000000000000008. PMID 24247114
- [Background] Scher JU, Ubeda C, Artacho A, Attur M, Isaac S, Reddy SM, Marmon S, Neimann A, Brusca S, Patel T, Manasson J, Pamer EG, Littman DR, Abramson SB. Decreased bacterial diversity characterizes the altered gut microbiota in patients with psoriatic arthritis, resembling dysbiosis in inflammatory bowel disease. Arthritis Rheumatol. 2015 Jan;67(1):128-39. doi: 10.1002/art.38892. PMID 25319745
- [Background] Zhang X, Zhang D, Jia H, Feng Q, Wang D, Liang D, Wu X, Li J, Tang L, Li Y, Lan Z, Chen B, Li Y, Zhong H, Xie H, Jie Z, Chen W, Tang S, Xu X, Wang X, Cai X, Liu S, Xia Y, Li J, Qiao X, Al-Aama JY, Chen H, Wang L, Wu QJ, Zhang F, Zheng W, Li Y, Zhang M, Luo G, Xue W, Xiao L, Li J, Chen W, Xu X, Yin Y, Yang H, Wang J, Kristiansen K, Liu L, Li T, Huang Q, Li Y, Wang J. The oral and gut microbiomes are perturbed in rheumatoid arthritis and partly normalized after treatment. Nat Med. 2015 Aug;21(8):895-905. doi: 10.1038/nm.3914. Epub 2015 Jul 27. PMID 26214836
- [Background] Yeoh N, Burton JP, Suppiah P, Reid G, Stebbings S. The role of the microbiome in rheumatic diseases. Curr Rheumatol Rep. 2013 Mar;15(3):314. doi: 10.1007/s11926-012-0314-y. PMID 23378145
- [Background] Scarpa R, Manguso F, D'Arienzo A, D'Armiento FP, Astarita C, Mazzacca G, Ayala F. Microscopic inflammatory changes in colon of patients with both active psoriasis and psoriatic arthritis without bowel symptoms. J Rheumatol. 2000 May;27(5):1241-6. PMID 10813294
- [Background] Van Praet L, Van den Bosch F, Mielants H, Elewaut D. Mucosal inflammation in spondylarthritides: past, present, and future. Curr Rheumatol Rep. 2011 Oct;13(5):409-15. doi: 10.1007/s11926-011-0198-2. PMID 21744132
- [Background] Lindqvist U, Kristjansson G, Pihl-Lundin I, Hagforsen E, Michaelsson G. Patients with psoriatic arthritis have an increased number of lymphocytes in the duodenal mucosa in comparison with patients with psoriasis vulgaris. J Rheumatol. 2006 May;33(5):924-7. Epub 2006 Mar 15. PMID 16541478
- [Background] Morgan XC, Huttenhower C. Meta'omic analytic techniques for studying the intestinal microbiome. Gastroenterology. 2014 May;146(6):1437-1448.e1. doi: 10.1053/j.gastro.2014.01.049. Epub 2014 Jan 28. PMID 24486053
- [Background] Klingberg E, Carlsten H, Hilme E, Hedberg M, Forsblad-d'Elia H. Calprotectin in ankylosing spondylitis--frequently elevated in feces, but normal in serum. Scand J Gastroenterol. 2012 Apr;47(4):435-44. doi: 10.3109/00365521.2011.648953. Epub 2012 Jan 10. PMID 22229862
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Smith MB, Kelly C, Alm EJ. Policy: How to regulate faecal transplants. Nature. 2014 Feb 20;506(7488):290-1. doi: 10.1038/506290a. No abstract available. PMID 24558658
- [Background] Toupin-April K, Barton J, Fraenkel L, Li L, Grandpierre V, Guillemin F, Rader T, Stacey D, Legare F, Jull J, Petkovic J, Scholte-Voshaar M, Welch V, Lyddiatt A, Hofstetter C, De Wit M, March L, Meade T, Christensen R, Gaujoux-Viala C, Suarez-Almazor ME, Boonen A, Pohl C, Martin R, Tugwell PS. Development of a Draft Core Set of Domains for Measuring Shared Decision Making in Osteoarthritis: An OMERACT Working Group on Shared Decision Making. J Rheumatol. 2015 Dec;42(12):2442-7. doi: 10.3899/jrheum.141205. Epub 2015 Apr 15. PMID 25877502
- [Background] Bruce B, Fries JF. The Health Assessment Questionnaire (HAQ). Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S14-8. PMID 16273780
- [Background] Faria JR, Aarao AR, Jimenez LM, Silva OH, Avelleira JC. Inter-rater concordance study of the PASI (Psoriasis Area and Severity Index). An Bras Dermatol. 2010 Sep-Oct;85(5):625-9. doi: 10.1590/s0365-05962010000500005. PMID 21152786
- [Background] Maksymowych WP, Mallon C, Morrow S, Shojania K, Olszynski WP, Wong RL, Sampalis J, Conner-Spady B. Development and validation of the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index. Ann Rheum Dis. 2009 Jun;68(6):948-53. doi: 10.1136/ard.2007.084244. Epub 2008 Jun 4. PMID 18524792
- [Derived] Kragsnaes MS, Jensen JRB, Nilsson AC, Malik MI, Munk HL, Pedersen JK, Horn HC, Kruhoffer M, Kristiansen K, Mullish BH, Marchesi JR, Kjeldsen J, Rottger R, Ellingsen T. Dynamics of inflammation-associated plasma proteins following faecal microbiota transplantation in patients with psoriatic arthritis and healthy controls: exploratory findings from the FLORA trial. RMD Open. 2024 Jan 30;10(1):e003750. doi: 10.1136/rmdopen-2023-003750. PMID 38296309
- [Derived] Parthasarathy R, Santiago F, McCluskey P, Kaakoush NO, Tedla N, Wakefield D. The microbiome in HLA-B27-associated disease: implications for acute anterior uveitis and recommendations for future studies. Trends Microbiol. 2023 Feb;31(2):142-158. doi: 10.1016/j.tim.2022.08.008. Epub 2022 Sep 1. PMID 36058784
- [Derived] Kragsnaes MS, Sodergren ST, Kjeldsen J, Horn HC, Munk HL, Pedersen JK, Klinkby CS, de Wit M, Ahlmark NG, Tjornhoj-Thomsen T, Ellingsen T. Experiences and perceptions of patients with psoriatic arthritis participating in a trial of faecal microbiota transplantation: a nested qualitative study. BMJ Open. 2021 Mar 8;11(3):e039471. doi: 10.1136/bmjopen-2020-039471. PMID 34006020
- [Derived] Kragsnaes MS, Kjeldsen J, Horn HC, Munk HL, Pedersen JK, Just SA, Ahlquist P, Pedersen FM, de Wit M, Moller S, Andersen V, Kristiansen K, Kinggaard Holm D, Holt HM, Christensen R, Ellingsen T. Safety and efficacy of faecal microbiota transplantation for active peripheral psoriatic arthritis: an exploratory randomised placebo-controlled trial. Ann Rheum Dis. 2021 Sep;80(9):1158-1167. doi: 10.1136/annrheumdis-2020-219511. Epub 2021 Apr 29. PMID 33926922
- [Derived] Kragsnaes MS, Kjeldsen J, Horn HC, Munk HL, Pedersen FM, Holt HM, Pedersen JK, Holm DK, Glerup H, Andersen V, Fredberg U, Kristiansen K, Christensen R, Ellingsen T. Efficacy and safety of faecal microbiota transplantation in patients with psoriatic arthritis: protocol for a 6-month, double-blind, randomised, placebo-controlled trial. BMJ Open. 2018 Apr 27;8(4):e019231. doi: 10.1136/bmjopen-2017-019231. PMID 29703851